CLINICAL TRIAL: NCT02733146
Title: Histones and Free-plasma DNA in the Days Following the Cardiac Arrest
Brief Title: Histones and Free-plasma DNA After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AU170878
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Heart Arrest; Hypothermia; Post Cardiac Arrest Syndrome
MeSH Terms: conditions — Heart Arrest; Hypothermia; Post-Cardiac Arrest Syndrome | interventions — Heart Arrest, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac arrest patients: Patients who has suffered a cardiac arrest
  Interventions: Other: cardiac arrest

INTERVENTIONS:
Other: cardiac arrest

SUMMARY:
To evaluate the significance of free-plasma deoxyribonucleic acid (DNA) and plasma histones in cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest of presumed cardiac cause
* Return of spontaneous circulation (ROSC)
* Glasgow Coma Score < 8
* Age > 18 years and < 80 years

Exclusion Criteria:

* >60 minutes from the circulatory collapse to ROSC
* Time interval > 4 hours from cardiac arrest to initiation of targeted temperature management
* Terminal illness
* Coagulation disorder
* Unwitnessed asystolia
* Cerebral performance category 3-4 before the cardiac arrest
* Severe persistent cardiogenic shock
* Pregnancy
* Persistent cardiogenic shock (systolic blood pressure < 80 despite inotropic treatment)
* New apoplexy or intracerebral hemorrhage
* Lack of consent from the relatives
* Lack of consent from the general practitioner
* Lack of consent from the patient if he/she wakes up and is relevant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest patients with a presumed cardiac origin, treated with targeted temperature management for 24 hours.
  For comparison; 20 healthy individuals were used.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Plasma histones | Approximate 24 hours after cardiac arrest
  The level of plasma histones
Free-plasma DNA | Approximate 24 hours after cardiac arrest
  The level of total free-plasma DNA

SECONDARY OUTCOMES:
Plasma histones | Approximate 48 hours and 72 hours after cardiac arrest
  The level of plasma histones
Free-plasma DNA | Approximate 48 hours and 72 hours after cardiac arrest
  The level of total free plasma DNA

OTHER OUTCOMES:
Simplified Acute Physiology Score (SAPS) score | Approximate 24 hours, 48 hours and 72 hours after cardiac arrest
Platelet count | Approximate 24 hours, 48 hours and 72 hours after cardiac arrest

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology and Intensive Care and Dept of Clinical Biochemistry, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No